CLINICAL TRIAL: NCT03049124
Title: Exercise for Adults Diagnosed With Rectal Cancer: A Feasibility Study
Brief Title: Exercise for Adults Diagnosed With Rectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to enroll participants into the study.
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Assistant Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RectalCaEx-JB-MV-KC
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Rectal Cancer
Keywords: Exercise; Feasibility trial; Cancer; Chemoradiation
MeSH Terms: conditions — Rectal Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Participants will be asked to complete a 12-week exercise intervention and all study assessments.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will engage in supervised exercise 3 times per week for 60-75 minutes/session for 12 weeks. Sessions will include a warm-up (aerobic activity less than < 60% of heart rate reserve), aerobic training (30 minutes of exercise at 60-75% of heart rate reserve, using cycle ergometers/treadmills), strength training (8 exercises; upper body, lower body, and core), and a cool-down (aerobic activity less than < 60% of heart rate reserve) component.

SUMMARY:
Currently, there is no clear indication if exercise is safe and if it confers health benefits for adults across the cancer trajectory (i.e., from diagnosis onward) for rectal cancer - a population who may have limited exercise tolerance and who may be at an increased risk for adverse events associated with exercise. In this prospective single-arm feasibility trial, we aim to examine the safety and feasibility of a 12-week exercise intervention for adults diagnosed with rectal cancer to inform the development of a large-scale randomized controlled trial that will assess the efficacy of exercise administered across the cancer trajectory for for rectal cancer. Adults who have been diagnosed with rectal cancer and are currently undergoing or have completed treatment (within the last five years) will be recruited over a 12-month period into a supervised exercise intervention consisting of aerobic and strength training to be done three times per week. Feasibility, safety, patient-reported outcomes, and physical tests will be performed pre-intervention and post-intervention. This study will provide data on the feasibility of an exercise intervention and will help determine if it is safe to progress with a large-scale randomized controlled trial to test the benefits of exercise for adults diagnosed with rectal cancer. It will also provide initial estimates of the parameters for patient-reported outcomes, which are required to calculate the sample size for the large-scale randomized controlled trial to ensure it is sufficiently powered.

The purpose of this prospective single-arm feasibility trial is to determine if a 12-week exercise intervention offered to adults diagnosed with rectal cancer surviviors is safe and feasible.

The specific objectives are to:

1. Test the feasibility and safety of a 12-week exercise intervention;
2. Obtain initial estimates of the parameters of the main outcomes to inform sample size calculations for the main study (i.e., means and standard deviations for patient-reported and physical outcomes);
3. Determine the opportune time in the cancer trajectory for rectal cancer to deliver a 12-week exercise intervention.

ELIGIBILITY:
Inclusion criteria are:

1. Men and women 18 to 85 years of age;
2. Diagnosed and/or completed treatment for stage I-III rectal cancer within the last 5 years;
3. Able to read/understand English or French;
4. Ambulatory;
5. Live <50km of the University of Ottawa;
6. Approval of healthcare provider to participate in the intervention.

Exclusion criteria are:

1. Congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, uncontrolled angina, uncontrolled arrhythmia, myocardial infarction, major heart surgery, stroke, or pulmonary embolus;
2. A diagnosis of hypertension or a resting blood pressure of 160/90 mmHg or higher (i.e., systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
3. The use of supplemental oxygen;
4. Severe arthritis (i.e., osteoarthritis or rheumatoid arthritis);
5. History of chest pain or severe shortness of breath either at rest or when engaging in physical activity;
6. Hip fracture, hip or knee replacement in the past 6 months;
7. Impairments requiring mobility aids;
8. Stage V cancer;
9. Prior cancer diagnosis, excluding non-melanoma skin cancer;
10. Participating in another exercise trial;
11. Unwilling/unable to give informed consent.

Of note, in addition to the exclusion criteria listed above, for individuals who are about to begin or are undergoing treatment healthcare providers will also employ clinical judgment concerning participant safety; that is, if the healthcare provider judges the patient to be at high risk for adverse events or medical complications if they participate in the intervention given their health status, they will not approach the patient to obtain permission for research personnel from the University of Ottawa to contact them.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | Through study completion, an average of 12 weeks
  The number of eligible participants who enrol in the study out of the number who are referred.
Retention Rates | Through study completion, an average of 12 weeks
  The number of participants completing the intervention and all scheduled assessments.
Adherence Rates | Through study completion, an average of 12 weeks
  The number of exercise sessions completed out of 36.
Number of Participants with Adverse Events | Through study completion, an average of 12 weeks
  The number of participants reporting or presenting adverse events (e.g., injury) that occurs as a result of participating in the exercise sessions and/or its assessments.

OTHER OUTCOMES:
Quality of Life: Functional Assessment of Cancer Therapy - Colorectal (Ward et al., 1999; Yost et al., 2005) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported quality of life from baseline to post-intervention.
Cognitive Functioning: Functional Assessment of Cancer Therapy - Cognitive Function (Wagner et al., 2004) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported cognitive function from baseline to post-intervention.
Symptoms of Fatigue: the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (Yellen et al., 1997) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported fatigue from baseline to post-intervention.
Affect: Positive and Negative Affect Schedule (Watson et al., 1988) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported affect from baseline to post-intervention.
Physical Activity Behaviour: Leisure Time Exercise Questionnaire (Godin & Shephard, 1985) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported physical activity (over the past 7 days) from baseline to post-intervention.
Resting Heart Rate: Heart Rate Monitor (Polar A300) | Baseline (week 0) and post-intervention (week 12)
  Change in resting heart rate from baseline to post-intervention.
Blood Pressure: Blood Pressure Monitor (HealthSmart Digital Blood Pressure Monitor) | Baseline (week 0) and post-intervention (week 12)
  Change in resting blood pressure from baseline to post-intervention.
Body Mass Index: Tanita Scale (TBF-310 GS) | Baseline (week 0) and post-intervention (week 12)
  Change in body mass index from baseline to post-intervention.
Aerobic Capacity: 6-Minute Walk Test (Canadian Society for Exercise Physiology, 2013; Irwin, 2012) | Baseline (week 0) and post-intervention (week 12)
  Change in aerobic capacity (i.e., total distance walked in 6 minutes) from baseline to post-intervention.
Musculoskeletal Strength: Combined Grip Strength Using a Handheld Dynamometer (Canadian Society for Exercise Physiology, 2013, 2013; Irwin, 2012) | Baseline (week 0) and post-intervention (week 12)
  Change in musculoskeletal strength (i.e., force exerted in kilograms on the handheld dynamometer) from baseline to post-intervention.
Socio-Demographic and Medical Information Questionnaire | Baseline (week 0)
  The socio-demographic and medical information collected will be used to describe the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brunet, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Society for Exercise Physiology. Canadian Society for Exercise Physiology - Physical activity training for health. Ottawa, ON: Canadian Society for Exercise Physiology, 2013.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Irwin ML. ACSM's guide to exercise and cancer survivorship. Champaign, IL: American College of Sports Medicine, 2012.
- [Background] Wagner LI, Cella D, Sweet J, Forrestal S. (2004). Chemotherapy-related cognitive deficits: development of the FACT-Cog instrument. Ann Behav Med, 27, S10.
- [Background] Ward WL, Hahn EA, Mo F, Hernandez L, Tulsky DS, Cella D. Reliability and validity of the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) quality of life instrument. Qual Life Res. 1999 May;8(3):181-95. doi: 10.1023/a:1008821826499. PMID 10472150
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Yost KJ, Cella D, Chawla A, Holmgren E, Eton DT, Ayanian JZ, West DW. Minimally important differences were estimated for the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) instrument using a combination of distribution- and anchor-based approaches. J Clin Epidemiol. 2005 Dec;58(12):1241-51. doi: 10.1016/j.jclinepi.2005.07.008. Epub 2005 Oct 13. PMID 16291468
- [Derived] Brunet J, Price J, Delluc C. An exercise trial for adults undergoing neoadjuvant chemoradiotherapy for rectal cancer proves not feasible: recommendations for future trials. Trials. 2021 Jan 6;22(1):26. doi: 10.1186/s13063-020-04958-z. PMID 33407782